CLINICAL TRIAL: NCT03810768
Title: Metabolomics Pilot Study on Postoperative Intensive Care Acquired Muscle Weakness (MIRACLE-I Study)
Brief Title: Metabolomics Study on Postoperative Intensive Care Acquired Muscle Weakness
Acronym: MIRACLE I
Status: Recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Helmholtz Zentrum München (Industry); Charite University, Berlin, Germany (Other); Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Stefan Schaller, MD, Principal Investigator, Medical University of Vienna
Other Study IDs: MIRACLE I
Record Dates: First submitted 2018-12-25; First posted 2019-01-22 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Metabolomics; Critical Care; Critical Illness; Critical Illness Myopathy; Critical Illness Polyneuropathy; Intensive Care (ICU) Myopathy; Muscle Weakness
Keywords: pilot trial; muscle biopsy; blood metabolome
MeSH Terms: conditions — Critical Illness; Polyneuropathies; Muscular Diseases; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood
  * Skeletal muscle biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intensive Care Patients: Postoperative high-risk patients who have been admitted to intensive care after surgery
- Operative Control patients: Elective operative patients where control blood samples and muscle ultrasound will be measured.

SUMMARY:
In this mono-center pilot trial, surgical patients who are at high risk to be admitted to intensive care will be screened and asked for participation. We are going to take blood and muscle samples at respecified time points to do metabolic, histological and molecular testing.

Aim of the study is to investigate (1) changes of the blood metabolome in patients with ICUAW (intensive care unit acquired weakness) and (2) identify metabolic components who are responsible for ICUAW or can be used as marker for ICUAW.

ELIGIBILITY:
Inclusion Criteria:

* invasive mechanically ventilated critically ill patient with expected intensive care unit stay > 3 days
* postoperative patient
* ≥ 18 years old
* American Society of Anesthesiology (ASA) classification ≥ III

Exclusion Criteria:

* moribund patient
* non-curative care (comfort care)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: mechanically ventilated postoperative high-risk patients who are admitted to intensive care
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolomics | a median of 14 days
  Blood Metabolome will be isolated from blood samples. All samples will be screened for influence of Intensive Care Unit Acquired Weakness (ICUAW) using mass spectrometry.

SECONDARY OUTCOMES:
Muscle histology | a median of 14 days
  Immunohistochemistry will be done in muscle samples. All samples will be screened for influence of Intensive Care Unit Acquired Weakness (ICUAW) and correlation with blood metabolome changes.
Phosphoproteomics | a median of 14 days
  Phosphoproteomics will be done in muscle samples using mass spectrometry. All samples will be screened for influence of Intensive Care Unit Acquired Weakness (ICUAW) and correlation with blood metabolome changes.

OTHER OUTCOMES:
Identify possible predictors of muscle wasting in the blood metabolome preoperatively | a median of 14 days
  Among the blood metabolome that will be measured, identify metabolites or combinations of metabolites whose high or low concentration(s) preoperatively associate(s) with the amount of muscle loss. These metabolites are candidate biomarkers that could be used to identify individuals at risk of large muscle wasting and may give further insights into the mechanisms of muscle wasting.
Identify possible predictors of muscle wasting in the blood metabolome at ICU admission | a median of 14 days
  Among the blood metabolome that will be measured, identify metabolites or combinations of metabolites whose high or low concentration(s) at ICU admission associate(s) with the amount of muscle loss. These metabolites are candidate biomarkers that could be used to identify individuals at risk of large muscle wasting and may give further insights into the mechanisms of muscle wasting.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Technical University of Munich; Hennig Wackerhage, PhD, Principal Investigator — Technical University of Munich
Locations (3):
- Medical University of Vienna, Vienna, Vienna, Austria
- Germany (2):
  - Klinikum rechts der Isar, School of Medicine, Technical University of Munich, Munich, Bavaria
  - Charité - Universitätsmedizin Berlin, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Undecided